CLINICAL TRIAL: NCT00167713
Title: Randomised, Double-Blind, Placebo Controlled Study of the Antipyretic Effect of Ibuprofen in Children With Uncomplicated Malaria
Brief Title: Treatment of Fever Due to Malaria With Ibuprofen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04/2003/IBU
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Fever
Keywords: Malaria; Fever; Ibuprofen; Gabon
MeSH Terms: conditions — Fever; Malaria | interventions — Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen

SUMMARY:
Drugs to treat fever are widely used in children with fever. But there is a controversy about the benefit of reducing fever in children with malaria. Ibuprofen is often used to treat malarial fever. This study evaluates the capacity of ibuprofen to reduce fever in malaria. The effect of ibuprofen on fever compared to only mechanical measures is investigated in children with malaria.

DETAILED DESCRIPTION:
Fever is the most apparent clinical manifestation of Plasmodium falciparum infection during the acute phase. The role of fever in defence against malaria or in other infectious diseases remains unclear. However, it has been shown that febrile temperatures inhibit the growth of P. falciparum in vitro.

Antipyretic drugs are commonly and widely used to treat malarial fever in endemic areas. There is however a controversy about the benefit of reducing fever in children with malaria. Data from Gabon have revealed that neither paracetamol, nor naproxen or metamizol - antipyretics often used in this area - had an effect on fever clearance time. Worryingly, paracetamol increased parasite-clearance times (i.e. inhibited clearance of parasites) and decreased significantly the production of oxygen radicals and tumour necrosis factor (TNF), mechanisms of the innate immune response, pivotal to combat infections.

Another antipyretic drug often used to treat malarial fever in endemic areas is ibuprofen. However, the rationale of its use and its capacity of reducing fever due to P. falciparum infections has never been proven in this area.

Comparison: The effect of ibuprofen plus mechanical fever "treatment" (continuous fanning, tepid sponging, and cooling blankets) is compared to mechanical treatment alone to treat fever in children with malaria.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated falciparum malaria
* Asexual parasitaemia between 20,000 and 200,000/µL
* Fever with temperature above 38 °C or history of fever during the preceding 24 hours
* Informed consent

Exclusion Criteria:

* Effective anti-malarial treatment for the present attack
* Antipyretic use within 6 hours of presentation
* Contraindications to the use of ibuprofen (history of asthma, dyspeptic symptoms, gastro-intestinal bleeding, or allergy to ibuprofen)
* Mixed plasmodial infection
* Haemoglobin < 7 g/dL
* Packed-cell volume < 20%
* White cell count > 16,000/L
* Platelet count < 40,000/µL
* Schizontaemia > 50/µL
* Impaired consciousness
* Convulsions or history of convulsions
* Concomitant diseases masking assessment of response

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2003-04; Study Completion 2004-01

PRIMARY OUTCOMES:
Fever clearance time
Fever time
Area under the fever curve

SECONDARY OUTCOMES:
Parasite clearance time
Adverse event during the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Michel A. Missinou, PhD, Principal Investigator — Albert Schweitzer Hospital
Locations (1):
- Medical research Unit, Lambaréné, Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Background] Kwiatkowski D. Febrile temperatures can synchronize the growth of Plasmodium falciparum in vitro. J Exp Med. 1989 Jan 1;169(1):357-61. doi: 10.1084/jem.169.1.357. PMID 2642531
- [Background] Long HY, Lell B, Dietz K, Kremsner PG. Plasmodium falciparum: in vitro growth inhibition by febrile temperatures. Parasitol Res. 2001 Jul;87(7):553-5. doi: 10.1007/s004360100374. PMID 11484852
- [Background] Kluger MJ. Drugs for childhood fever. Lancet. 1992 Jan 4;339(8784):70. No abstract available. PMID 1346006
- [Background] Brandts CH, Ndjave M, Graninger W, Kremsner PG. Effect of paracetamol on parasite clearance time in Plasmodium falciparum malaria. Lancet. 1997 Sep 6;350(9079):704-9. doi: 10.1016/S0140-6736(97)02255-1. PMID 9291905
- [Background] Lell B, Sovric M, Schmid D, Luckner D, Herbich K, Long HY, Graninger W, Kremsner PG. Effect of antipyretic drugs in children with malaria. Clin Infect Dis. 2001 Mar 1;32(5):838-41. doi: 10.1086/319217. Epub 2001 Feb 23. PMID 11229858
- [Background] Krishna S, Pukrittayakamee S, Supanaranond W, ter Kuile F, Ruprah M, Sura T, White NJ. Fever in uncomplicated Plasmodium falciparum malaria: randomized double-'blind' comparison of ibuprofen and paracetamol treatment. Trans R Soc Trop Med Hyg. 1995 Sep-Oct;89(5):507-9. doi: 10.1016/0035-9203(95)90087-x. PMID 8560525
- [Background] Nwanyanwu OC, Ziba C, Kazembe PN. Paracetamol and ibuprofen for treatment of fever in Malawian children aged less than five years. Trans R Soc Trop Med Hyg. 1999 Jan-Feb;93(1):84. doi: 10.1016/s0035-9203(99)90191-8. No abstract available. PMID 10492798
- [Derived] Matsiegui PB, Missinou MA, Necek M, Mavoungou E, Issifou S, Lell B, Kremsner PG. Antipyretic effect of ibuprofen in Gabonese children with uncomplicated falciparum malaria: a randomized, double-blind, placebo-controlled trial. Malar J. 2008 May 26;7:91. doi: 10.1186/1475-2875-7-91. PMID 18503714
- See also: General information on malaria at the website of the Malaria Foundation International — http://www.malaria.org
- See also: Homepage of the Medical Research Unit, Lambaréné — http://www.lambarene.org